CLINICAL TRIAL: NCT03533010
Title: Preventing Curve Progression and the Need for Bracing in Early Diagnosed Adolescent Idiopathic Scoliosis Using Calcium Plus Vitamin D Supplementation - A Randomized Double-blinded Placebo-controlled Trial
Brief Title: Preventing Curve Progression and the Need for Bracing in Adolescent Idiopathic Scoliosis With Calcium + Vitamin D Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tsz-ping Lam, Associate Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CalE_Protocol_V04
Record Dates: First submitted 2018-04-30; First posted 2018-05-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Scoliosis; Spinal Curvatures; Spinal Diseases; Bone Health; Vitamin D
Keywords: Adolescent Idiopathic Scoliosis; Bone Health; Treatment; Vitamin D; Calcium
MeSH Terms: conditions — Scoliosis; Spinal Curvatures; Spinal Diseases | interventions — Calcium; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ca500mg + VitD800IU (Active Comparator): Daily Supplementation with 500mg Calcium plus 800IU Vitamin D3
  Interventions: Dietary Supplement: Ca500mg; Dietary Supplement: VitD800IU
- Placebo (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ca500mg — subjects receive a daily dose of 500mg elemental calcium
  Other Names: Calcium 500mg
  Arms: Ca500mg + VitD800IU
Dietary Supplement: VitD800IU — subjects receive a daily dose of 800IU VitD3
  Other Names: Vitamin D3 800IU
  Arms: Ca500mg + VitD800IU
Other: Placebo — subjects receive placebo tablet
  Arms: Placebo

SUMMARY:
There is an association between adolescent idiopathic scoliosis (AIS) and low bone mass which has been reported to be a significant prognostic factor for curve progression. Given that dietary calcium (Ca) intake and serum Vit-D levels were also low in AIS, we therefore propose a randomized double-blinded placebo-controlled trial to evaluate if daily [500mg Ca + 800 IU Vit-D] can improve bone health and prevent curve progression in AIS. Immature AIS girls with Cobb angle 10-20 degrees will be randomized either to the Treatment or Placebo group with 3-year of treatment. The main outcome measures for evaluation for those who have completed the 3-year treatment and have reached skeletal maturity at the end of 3-year treatment include: (1) percentage of patients with increase in Cobb angle≥6 degrees and (2) percentage of patients who require bracing. Bone measurements using advanced image acquisition technology(HR-pQCT) to assess bone health will also be evaluated.

DETAILED DESCRIPTION:
This study investigates if calcium (Ca) plus Vitamin D (Vit-D) supplementation can prevent curve progression and improve bone health in early Adolescent Idiopathic Scoliosis (AIS) during pubertal growth.

AIS is a prevalent three-dimensional spinal deformity mainly affecting girls at puberty. It can lead to serious complications including spine degeneration, cardiopulmonary compromise, grossly deformed torso and psychosocial disorders. Current treatments are far from being satisfactory, with bracing being lengthy and physically demanding and surgery being a major invasive procedure.

There is an association between AIS and low bone mass which has been reported to be a significant prognostic factor for curve progression. Given that dietary calcium intake and serum Vit-D levels were also low in AIS, we therefore propose a randomized double-blinded placebo-controlled trial to evaluate if daily [500mg Ca + 800 IU Vit-D] can improve bone health and prevent curve progression. Immature AIS girls with Cobb angle 10-20 degrees will be randomized either to the Treatment or Placebo group with 3-year of treatment. The main outcome measures for evaluation for those who have completed the 3-year treatment and have reached skeletal maturity at the end of 3-year treatment include: (1) percentage of patients with increase in Cobb angle≥6 degrees and (2) percentage of patients who require bracing. Bone measurements using advanced image acquisition technology (HR-pQCT) to assess bone health will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. girls with diagnosis of AIS confirmed after detailed clinical and radiological assessment and
2. between 10 to 14 years old and
3. Risser between 0 to 2 and
4. pre-menarche or < 1 year post-menarche and
5. Cobb angle between 10° to 20 ° and
6. no prior bracing or other treatment for scoliosis and
7. no prior treatment for bone health

Exclusion Criteria:

1. scoliosis with any known etiology such as congenital scoliosis, neuromuscular scoliosis, scoliosis of metabolic etiology, scoliosis with skeletal dysplasia or
2. patients with known endocrine and connective tissue abnormalities, or
3. patients with eating disorders or gastrointestinal malabsorption disorders or any disorders that are known to affect calcium or bone metabolism or
4. prior treatment for bone health before being recruited into the study or
5. patient currently taking medication that affects bone metabolism eg steroid or
6. patient with contra-indications for calcium and Vit-D supplementation:

   1. history of hypersensitivity to the active or placebo tablets
   2. history of renal diseases and renal calculi (nephrolithiasis)
   3. diseases and/or conditions resulting in hypercalcaemia and/or hypercalciuria
   4. hypervitaminosis D

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 199 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Curve progression (Cobb) | 3 years
  Percentage of patients with increase in Cobb angle ≥ 6 degrees
Curve progression (Bracing) | 3 years
  Percentage of patients who require bracing

SECONDARY OUTCOMES:
Bone health (BMD) | 3 years
  Improvement in areal bone mineral density measured with Dual-energy X-ray absorptiometry
Bone health (bone quality) | 3 years
  Improvement in bone quality measured with High-resolution peripheral quantitative computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Ping Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No